CLINICAL TRIAL: NCT06247397
Title: Effect of HIgh-flow Therapy in Long-term Oxygen Therapy (HILOT): A Multicenter, Registry-based, Randomized Clinical Trial
Brief Title: Effect of HIgh-flow Therapy in Long-term Oxygen Therapy
Acronym: HILOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Uppsala University Hospital (Other); Region Stockholm (Other Government); Region Örebro County (Other); Blekinge County Council Hospital (Other); Blekinge Institute of Technology (Other); Lund University (Other); Region Östergötland (Other); Vastra Gotaland Region (Other Government); Region Västerbotten (Other Government); Landstinget i Värmland (Other); ResMed (Industry); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Magnus Ekström, Associate Professor, Senior Lecturer, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HILOT
Record Dates: First submitted 2024-01-17; First posted 2024-02-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Interstitial Lung Disease; Chronic Respiratory Failure With Hypoxia
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-flow oxygen therapy (Experimental): Intervention arm
  Interventions: Device: Added high-flow oxygen therapy
- Low-flow oxygen therapy (Active Comparator): Comparison arm
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Added high-flow oxygen therapy — Added high-flow oxygen therapy using the device Lumis HFT during nighttime and at the patient's discretion daytime, with the usual care (low-flow oxygen therapy) the rest of the time.
  Arms: High-flow oxygen therapy
Other: Standard care — Standard care with low-flow oxygen therapy in accordance with clinical routine.
  Arms: Low-flow oxygen therapy

SUMMARY:
This is a registry-based, randomized, controlled clinical trial of the effect of added high-flow oxygen therapy (using the device Lumis HFT) during one year in people with long-term oxygen therapy (LTOT) for chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD).

DETAILED DESCRIPTION:
This is a registry-based, randomized, controlled clinical trial of patients with LTOT for COPD or ILD recruited using the Swedish National Registry for Respiratory Failure (Swedevox) in collaboration with a research network within the Swedish Respiratory Society. The trial evaluates the effect of added high-flow oxygen therapy nighttime to the regular low-flow oxygen therapy compared with regular low-flow oxygen therapy alone up to one year.

The purpose of this project is to improve evidence-based treatment of people with chronic respiratory failure, currently about 2000 patients annually in Sweden, who have high risk of adverse events and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Ongoing LTOT: prescribed for at least 15 hours per day; and since at least 28 days as registered in Swedevox
* COPD or ILD as main underlying reason for LTOT
* Oxygen concentrator as stationary oxygen source in the home including night-time
* Body mass index (BMI) < 35 kg/m2

Exclusion Criteria:

* Current or previous treatment with home HFOT
* Current treatment with home mechanical ventilation
* Current treatment with home CPAP
* Hospitalized during the last 2 weeks
* Current smoking or contact with flames
* Self-reported average use of the LTOT < 15h per day (24 hours)
* PaCO2 (breathing air at rest) > 8 kPa
* Strong clinical suspicion of obstructive sleep apnea (OSA) or obesity-related hypoventilation syndrome (OHS) (as judged by the responsible staff)
* Inability to participate in the study procedures (as judged by the staff)
* Not eligible for continuing LTOT due to other reason (as judged by the staff)
* Expected survival less than 3 months (as judged by the staff)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to first hospitalization or death from all causes | 1 year
  Time to first hospitalization or death from all causes during 1 year after randomization in people with COPD (assessed using nationwide registry data)

SECONDARY OUTCOMES:
Time to first all-cause hospitalization or all-cause death | 1 year
  Time to first all-cause hospitalization or all-cause death in people with ILD (assessed using nationwide registry data)
Rate of hospitalizations or death from all causes | 1 year
  Rate of hospitalizations or death from all causes assessed using nationwide registry data
Hospitalization rate from all causes | 1 year
  Hospitalization rate from all causes assessed using nationwide registry data
Hospitalization rate from respiratory disease | 1 year
  Hospitalization rate from respiratory disease assessed using nationwide registry data
Number of hospitalized days | 1 year
  Number of hospitalized days from all-causes, respiratory and cardiovascular disease using nationwide registry data
Hospitalization rate from cardiovascular disease | 1 year
  Hospitalization rate from cardiovascular disease assessed using nationwide registry data
Number of admissions to intensive care unit (ICU) | 1 year
  Number of admissions to ICU assessed using nationwide registry data
Number of days in ICU | 1 year
  Number of days in ICU assessed using nationwide registry data
Mortality rate from all causes | 1 year
  The mortality rate from all causes assessed using nationwide registry data
Mortality rate from respiratory disease | 1 year
  The mortality rate from respiratory disease assessed using nationwide registry data
Mortality rate from cardiovascular disease | 1 year
  The mortality rate from cardiovascular disease assessed using nationwide registry data
Time to first exacerbation | 1 year
  Time to first exacerbation after randomisation, defined as time to first dispensed antibiotics and/or oral corticosteroids, ED-visit or hospitalization for exacerbation assessed using self-reported and registry data
Number of exacerbations | 1 year
  Number of exacerbations of all severity assessed using self-reported and registry data
Incidence of cardiovascular disease | 1 year
  Incidence of cardiovascular disease assessed using nationwide registry data
Need for home mechanical ventilation | 1 year
  Need for starting home mechanical ventilation assessed using nationwide registry data
Rate of withdrawal of long-term oxygen therapy | 1 year
  Rate of withdrawal of long-term oxygen therapy assessed using nationwide registry data
Adverse events | 3 and 12 months
  Self-reported adverse events since study start assessed using a postal questionnaire.
Primary care utilization | 1 year
  Self-reported number of primary care contacts since the start of the study assessed using a postal questionnaire.
Health-related quality of life | 3 and 12 months
  Self-reported health-related quality of life assessed using the EuroQol Five Dimensions - Five Levels (EQ5D-5L) questionnaire.
Health status | 3 and 12 months
  Self-reported health status assessed using the and the COPD Assessment Test (CAT) questionnaire.
Breathlessness at exertion | 3 and 12 months
  Self-reported exertional breathlessness assessed using the Dyspnoea Exertion Scale (DES) questionnaire.
Breathlessness | 3 and 12 months
  Self-reported breathlessness assessed using the Dyspnea-12 questionnaire.
Sleep quality | 3 and 12 months
  Self-reported sleep quality assessed using the modified Basic Nordic Sleep Questionnaire.
Physical activity | 3 and 12 months
  Self-reported level of physical activity assessed using the modified Grimby-Frändin questionnaire.
Change in health status | 3 and 12 months
  Self-reported change in perceived health status assessed using the Global Impression of Change (GIC) scale.
Nasal symptoms | 3 and 12 months
  Self-reported nasal symptoms assessed using the modified Björklund questionnaire.

OTHER OUTCOMES:
Patient preference for continuing the treatment | 3 and 12 months
  Patients' self-reported patient preference for continuing the treatment assessed using postal questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ekström, MD, PhD, Principal Investigator — Skane University Hospital
Locations (2):
- Sweden (2):
  - Research Unit, Blekinge University of Technology, Karlskrona, Blekinge County
  - Department of Heart, Lung and Clinical Physiology, Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No
IPD cannot be shared due to restrictions in the current ethical approval. Pseudonymized IPD can be shared upon reasonable request and separate ethical approval.

REFERENCES:
- [Derived] Sundh J, Ljunggren M, Palm A, Lindberg E, Lavergne F, Weinreich UM, Ahmadi Z, Ekstrom M; HILOT Collaboration Group. Effect of HIgh-Flow Therapy in Long-Term Oxygen Therapy (HILOT): study protocol for a multicentre, registry-based, randomised clinical trial. Trials. 2026 Feb 4. doi: 10.1186/s13063-026-09488-8. Online ahead of print. PMID 41634827